CLINICAL TRIAL: NCT00004784
Title: Phase III Randomized Study of Ursodiol With Vs Without Methotrexate for Primary Biliary Cirrhosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Texas (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/11873; UTSMC-29205400
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Liver Cirrhosis, Biliary
Keywords: cirrhosis; gastrointestinal disorders; primary biliary cirrhosis; rare disease
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Fibrosis; Gastrointestinal Diseases; Rare Diseases | interventions — Methotrexate; Ursodeoxycholic Acid

INTERVENTIONS:
Drug: methotrexate
Drug: ursodiol

SUMMARY:
OBJECTIVES: I. Compare the effects of ursodiol (ursodeoxycholic acid), with and without methotrexate, on pruritus, incapacitation index, and serum markers of activity and severity in patients with primary biliary cirrhosis.

II. Compare the effects of these regimens on the development of ascites, encephalopathy, varices (or bleeding from pre-existing varices), histologic liver changes, transplantation, and survival.

III. Compare the toxicity and safety of each regimen.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double-blind study. Patients are stratified by participating institution and Ludwig histologic stage.

All patients are treated with ursodiol (ursodeoxycholic acid, UDCA) for 6 months. If entry criteria continue to be met, patients are randomly assigned to UDCA/methotrexate or UDCA/placebo.

Combination therapy continues for at least 5 years.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- The following criteria must be met prior to study entry and ursodiol treatment: Bilirubin less than 3 mg/dL Alkaline phosphatase at least 1.5 times normal limits Albumin at least 3 g/dL The following criteria must be met prior to randomization to Arms I and II: Primary biliary cirrhosis (PBC), i.e.: Cholestatic liver disease for at least 6 months prior to randomization Liver biopsy compatible with PBC within 6 months prior to randomization No biliary obstruction on ultrasound, computerized tomography, or cholangiography The following exclude: Asymptomatic and stage I liver histology (Ludwig classification) Hepatic encephalopathy Ascites Variceal bleeding No liver disease of other etiology, e.g.: Chronic hepatitis B or C Autoimmune chronic active hepatitis Alcoholic liver disease Sclerosing cholangitis Drug-induced liver disease Symptomatic or obstructive gallstones --Prior/Concurrent Therapy-- At least 6 months since the following immunosuppressives: Cyclosporine Tacrolimus Methotrexate At least 3 months since other immunosuppressives, e.g.: Azathioprine Chlorambucil Colchicine Corticosteroids Penicillamine At least 3 months since rifampin --Patient Characteristics-- Life expectancy: No major illness limiting life span Hematopoietic: WBC at least 2500/mm3 Absolute granulocyte count at least 1500/mm3 Platelet count at least 80,000/mm3 Hepatic: See Disease Characteristics Renal: Creatinine clearance at least 60 mL/min Pulmonary: No diffusion capacity or vital capacity less than 50% of predicted Other: Antimitochondrial antibody positive HIV antibody negative No alcoholism within the past 2 years No epilepsy requiring phenytoin No malignancy within the past 5 years other than skin cancer No pregnant women Adequate contraception required of fertile patients

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315
Dates: Start 1994-01

CONTACTS AND LOCATIONS:
Overall Officials: Burton Combes, Study Chair — University of Texas